CLINICAL TRIAL: NCT04858490
Title: Remote Treatment of Alcohol Withdrawal: A Pilot Study
Brief Title: Remote Treatment of Alcohol Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137/2020
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Withdrawal
Keywords: Withdrawal Management; Telemedicine; Alcohol Withdrawal; Alcohol Withdrawal Management; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptom-triggered diazepam treatment (Experimental): Participants will be treated for a period of 3 days using a symptom-triggered withdrawal management protocol delivered over telemedicine. Participants who score 10 or above on the modified CIWA-Ar will be advised to take a specific dose of diazepam (either 10 or 20mg, at the clinician's discretion). Participants will be reassessed regularly over the 3-day period.
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam — Symptom-triggered diazepam treatment: 10 or 20mg, at the clinician's discretion
  Other Names: Valium

SUMMARY:
This study will evaluate the feasibility of delivering symptom-triggered alcohol withdrawal management by telemedicine and determine whether this intervention is satisfactory to patients.

DETAILED DESCRIPTION:
This single-arm pilot feasibility study will recruit actively drinking participants with a history of alcohol withdrawal in order to provide remotely monitored symptom-triggered alcohol withdrawal treatment using telemedicine. Participants will initially complete a screening and eligibility visit. If eligible, participants will then be scheduled for 3-day remote withdrawal management (which can be extended by 1-2 days if medically indicated). During remote withdrawal management, participants will receive symptom-triggered diazepam treatment using a modified version of the Clinical Institute Withdrawal Assessment for Alcohol Scale, revised (CIWA-Ar). Within one week following termination of withdrawal treatment, participants will be scheduled for a remote follow up visit in which they will complete patient satisfaction questionnaires and will be offered weekly counselling sessions and anticraving medication to prevent relapse to alcohol use. Approximately 30 days following treatment initiation, relapse to alcohol use will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Are actively using alcohol
* Previously met Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) B criteria for alcohol withdrawal
* Aim to achieve at least 30 days of abstinence as a treatment goal following initiation of remote alcohol withdrawal management
* Are able to provide informed consent in English.
* Reside or are able to stay at an address within 2-hours travelling distance from the Centre for Addiction and Mental Health for the entire duration of the remote withdrawal procedure
* Are enrolled in the Ontario Health Insurance Plan (OHIP)

Exclusion Criteria:

* History of complicated withdrawal including withdrawal seizures, hallucinosis, or delirium
* Positive UDS for sedatives or opioids, currently prescribed sedatives or opioids, or diagnosis of sedative-hypnotic or opioid use disorder within the past year (based on assessment). Individuals prescribed low doses of benzodiazepines (e.g. lorazepam 1mg PO daily) or with a positive urine benzodiazepine screen that is not thought to be due to benzodiazepine misuse may be permitted to proceed with the study at the discretion of the study physician.
* Severe medical or psychiatric comorbidity that would prevent safe participation in the study
* Contraindications to the safe use of diazepam including: known hypersensitivity to diazepam severe respiratory insufficiency, severe hepatic insufficiency, sleep apnea syndrome, acute narrow-angle glaucoma, and myasthenia gravis. Individuals with sleep apnea may be permitted to proceed with the study at the discretion of the study physician.
* Active withdrawal symptoms (CIWA-Ar > 12) at the time of the eligibility assessment
* Active suicidal ideation at the time of eligibility assessment
* Positive urine pregnancy test, actively breastfeeding, or planning to become pregnant or breastfeed during the study period
* Lack of stable housing
* Enrollment in another study that conflicts with the procedures or scientific integrity of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Retention in treatment | 3-5 day treatment period
  Retention in treatment, as measured by the percentage of participants who complete the entire 3-day remote withdrawal management protocol.
Transfer to a higher level of care | 3-5 day treatment period
  Transfer to a higher level of care, as measured by the percentage of participants sent to the emergency room due to complications, need for intensive monitoring, or acute intoxication.

SECONDARY OUTCOMES:
Patient satisfaction with the treatment protocol | Measured within 1 week of completing the remote withdrawal procedure
  Satisfaction with the overall treatment protocol, measured with the Client Satisfaction Questionnaire-8 (minimum score = 8; maximum score = 32; higher score indicates greater client satisfaction).
Patient satisfaction with the telemedicine platform | Measured within 1 week of completing the remote withdrawal procedure
  Satisfaction with the telemedicine platform, measured with a modified version of the Telehealth Satisfaction Scale (minimum score = 12; maximum score = 48; higher score indicates greater satisfaction with the telemedicine platform).
Duration of active withdrawal treatment | 3-5 day treatment period
  Duration of active withdrawal treatment, as measured by the number of days that patients received diazepam among patients who received benzodiazepines.
Requirement of benzodiazepines | 3-5 day treatment period
  Benzodiazepines requirement, as measured by the percentage of participants requiring benzodiazepine treatment.
Diazepam dose | 3-5 day treatment period
  Diazepam dose, as measured by the average dose of diazepam required to control symptoms among patients who received diazepam.
Withdrawal severity | 3-5 day treatment period
  Withdrawal severity, as measured by the average peak Clinical Institute Withdrawal Assessment for Alcohol Scale, revised score measured over the treatment period (minimum score = 0; maximum score = 67; higher score indicates greater withdrawal severity).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sloan, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No